CLINICAL TRIAL: NCT03724708
Title: Comparing Expulsion Rates When Using "Hang Up" Intrauterine Device Insertion Technique to Postplacental and Postpartum Insertion
Brief Title: Comparing Expulsion Rates for Different Intrauterine Device Insertion Techniques
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Ahmed M.Kamel, Asst. Professor of obstetrics and gynecology, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: A10102018
Record Dates: First submitted 2018-10-16; First posted 2018-10-30 (Actual); Last update posted 2018-12-04 (Actual); Status verified 2018-12

CONDITIONS: IUD Insertion Complication; IUD; Complications, Infection or Inflammation
Keywords: IUD expulsion; hang up technique; postpartum insertion
MeSH Terms: conditions — Infections; Inflammation

STUDY DESIGN:
Intervention Model Description: randomized controlled trial
Who Masked: Participant
Masking Description: randomised computer generated table and closed envelope system
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Hang up technique (Experimental): where the enrolled patients will have the IUD applied in the middle of the uterine cavity and then attached to the fundus of the uterus by an absorbable suture "Hang up technique"
  Interventions: Device: IUD
- Postpartum insertion (Active Comparator): will include patients where IUD will be inserted after 6 weeks post-partum.
  Interventions: Device: IUD
- Control (Active Comparator): will serve as our control group where the enrolled patients will have the IUD just applied into the middle of the uterine cavity at the level of the fundus without attachment
  Interventions: Device: IUD

INTERVENTIONS:
Device: IUD — IUD insertion

SUMMARY:
the investigators are trying to determine if this method of intrauterine device (IUD) insertion "hang up technique" has less expulsion rates than 6 week insertion or immediate post-placental insertion.

DETAILED DESCRIPTION:
This prospective multi-center clinical trial will be conducted at the Kasr Alainy maternity hospital, and AL-Zahra university hospital after approval from both ethics committees was obtained (OBGYN Scientific & ethics committee and Al-Zahra ethics committee). The study will enroll pregnant women attending the antenatal care clinic who have been scheduled for elective cesarean section after obtaining a signed informed consent from all participants.

The enrolled participants will be divided into 3 groups:

* Group A: will serve as our experimental group where the enrolled patients will have the IUD applied in the middle of the uterine cavity and then attached to the fundus of the uterus by an absorbable suture "Hang up technique" (Tjahjanto & Haryuni, 2014)
* Group B: will serve as our active comparator and will include patients where IUD will be inserted after 6 weeks post-partum.
* Group C: will serve as our control group where the enrolled patients will have the IUD just applied into the middle of the uterine cavity at the level of the fundus without attachment.

Randomization will be done by a computer-generated randomization table, and assignment into the various groups will be done by a sealed opaque envelope system which will be opened by the circulating nurse in the operating room during cesarean section.

In both groups A and C, a Copper T-380 IUD (TCU 380 A with safe load PREGNA INTERNATIONAL LTD® manufactured by PREGNA® - India) was placed in the middle of the uterine cavity, and the threads was passed through the cervix after dilatation by one finger.

In group (A) Hang up technique will be done with the same technique of a previous study done by Tjahjanto and Haryuni in 2014, but by using 2-0 Polyglactin 910 undyed braided absorbable suture with a straight needle "KS 60mm reverse cutting" (VICRYL RAPIDE™ ETHICON®). The needle will be inserted perpendicularly from the outside the uterus to penetrate the median of the fundus wall to get into the uterine cavity. Once the surgical thread entered the uterine cavity, the needle is clamped with rings forceps and pulled out through the lower uterine segment incision. Subsequently, an anchor knot is made on the crossing arm so that the IUD is balanced and hanging flexibly on the wall of the fundus. The IUD string is then cut in the middle of the long thread. Using ring forceps for clamping the IUD, it is inserted into the uterine cavity while simultaneously pulling the surgical thread out of the uterus so that the IUDs horizontal arm is touching the uterine fundus. The position of IUD remains suspended by the thread. Then, a knot is made on the outer surface of the uterus so the IUD will be fixed and hangs from the fundus (Tjahjanto & Haryuni, 2014) The patients will be evaluated for postpartum hemorrhage and fever 24 hours following the surgery. Patients will be re-evaluated 6 weeks, 3 and 6months postpartum for vaginal bleeding (irregular bleeding and menorrhagia), vaginitis (smelly odor, discharge) PID (fever, ovarian abscess, hydro/pyo-salpinx).

Patients will also be re- evaluated by trans-vaginal ultrasound (US) to assess the position of IUD inside uterine cavity at 24hours, also at 6 weeks, 3and 6 months post-operative. Expulsion is defined when the IUD is not seen inside the uterine cavity by US and fundal displacement is noted when distance between transverse limb of IUD and fundus more than 20mm.

If the acceptor does not arrive on time, they will be invoked by a call. If they cannot be contacted or found until the end of the study they will be considered as loss of follow-up.

sample size: the investigators are planning a study of independent cases and controls with 1 control(s) per case. Prior data indicate that the probability of exposure among controls is 0.044. If the true probability of exposure among cases is 0. 24 (Chen et al, 2010). We will need to study 49 case patients and 49 control patients to be able to reject the null hypothesis that the exposure rates for case and controls are equal with probability (power) 0.8. The Type I error probability associated with this test of this null hypothesis is 0.05. we will increase the number of participants to 54 in each group (10%) to allow for drop outs.

ELIGIBILITY:
Inclusion Criteria:

* Full term patients (≥ 37 weeks gestation).
* Singleton pregnancy.
* Elective cesarean section for an uncomplicated pregnancy.
* Healthy uterine cavity (no fibroid and no congenital anomaly) (Previously documented by history taking and/or ultrasound before pregnancy, and to be re-confirmed intraoperative).

Exclusion Criteria:

* Preterm labor.
* Uterine fibroid distorting uterine cavity.
* History suggestive of previous pelvic inflammatory disease (Fever due to vaginal infection, ovarian abscess, repeated offensive vaginal infection, hydro/pyo-salpinx) 2
* Rupture of membrane more than 12 hours.
* Multi-fetal pregnancy
* Placenta previa.
* Previous uterine surgery other than CS
* Documented congenital uterine anomalies intraoperative.
* History of IUD insertion before this pregnancy with side effects like "bleeding, ectopic pregnancy, expulsion, pelvic inflammatory disease"
* Uterine atony after delivery.

Ages: 22 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 162 (Estimated)
Dates: Start 2018-12-02 (Actual); Primary Completion 2019-08 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Expulsion rates | 6months
  IUD expulsion among the 3 groups at different intervals 24hours, 6 weeks, 3 and 6months postpartum

SECONDARY OUTCOMES:
Temperature | 24 hours
  postpartum fever (38 degrees celsius or above)
Irregular bleeding | 6 months.
  defined as irregular bleeding and menorrhagia discovered at 6 weeks, 3 and 6months postpartum
Vaginitis | 6 months
  Defined as smelly odor, discharge diagnosed at 6 weeks, 3 and 6months postpartum
postpartum hemorrhage | 24 hours
  Defined as heavy bleeding after delivery diagnosed in the first 24 hours after labor

CONTACTS AND LOCATIONS:
Overall Officials: Mamoud Soliman, M.D., Principal Investigator — Lecturer of obstetrics and gynecology
Locations (1):
- obstetrics and gynecology department, Kasr Alainy hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Goldstuck ND, Wildemeersch D. Role of uterine forces in intrauterine device embedment, perforation, and expulsion. Int J Womens Health. 2014 Aug 7;6:735-44. doi: 10.2147/IJWH.S63167. eCollection 2014. PMID 25143756
- [Background] Chen BA, Reeves MF, Hayes JL, Hohmann HL, Perriera LK, Creinin MD. Postplacental or delayed insertion of the levonorgestrel intrauterine device after vaginal delivery: a randomized controlled trial. Obstet Gynecol. 2010 Nov;116(5):1079-87. doi: 10.1097/AOG.0b013e3181f73fac. PMID 20966692
- [Background] Tjahjanto H, Haryuni IT. Hang-up IUD, new technique for suturing CuT-380A IUD to uterine fundus in immediate postplacental insertion during cesarean delivery: twelve months follow up. Indones J Obstet Ginecol. 2014;2-31:132-139.